CLINICAL TRIAL: NCT03889717
Title: A Randomized Controlled Trial Comparing Two Regimens of Vitamin D Supplementation in Preterm Neonates
Brief Title: Comparison of Two Different Doses of Vitamin D in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Jamal Abd elmoez abd elmegeed Basta, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPTL
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteopenia of Prematurity
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: after randomization ,two different groups of premature neonates are enrolled in the study baseline calcium,phosphorus and alp and vitamin D withdrawn at the 1st 48 hrs, then neonates started to administer vitamin D drops after they reached 100 cc per kg per day until they complete 40th week gestational age .follow up labs will be done at this age to determine which dose is better in vitamin d deficiency prevention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 400 iu (Experimental): neonates who will receive vitamin d dose at 400 iu per day
  Interventions: Dietary Supplement: vitamin D
- 1000 iu (Active Comparator): neonates who will receive vitamin d dose 1000 iu per day
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — vitamin d drops will be given daily to the 2 groups of neonates ( 1st group will be given 400 iu /day and 2nd group will be given 1000 iu per day ) when they reach 100 cc per kg enteral feeding .. until they reach 40 weeks gestational age

SUMMARY:
randomized clinical trial comparing two different doses of vitamin d supplementation in preterm infants

DETAILED DESCRIPTION:
after randomization each group of preterm neonates (28-32) weeks consisting of 40 neonates

within 48 hrs of birth baseline ca.phosphorus, alkaline phosphatase and vitamin D level were withdrawn from each neonate

then babies started to take oral vitamin d in different doses (400 IU /day in the 1st group and 1000 iu per day in the 2nd group) after they reach 100 cc per kg per day enteral feeding

after they complete 40th week gestational age the investigators repeat the labs again ( serum ca, phosphorus,alp and vitamin D and compare the rate of rise in vitamin D and calcium

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants delivered at a gestational age ≤ 32 weeks
* Birth weight ≤1500 kg

Exclusion Criteria:

* Neonates with major congenital anomalies,
* maternal condition or medications likely to influence vitamin D or calcium metabolism
* neonates not receiving 100 ml/ kg / day of enteral feeds by 14 days of life

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the level of serum 25 hydroxy vitamin D between the two groups of newborns. 2- Detect vitamin D deficiency among both groups. | 1 month
  measurement of the level after supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided